CLINICAL TRIAL: NCT04419792
Title: 'A Profile of Physical Performance Variables in an Out-patient Adult Population With Narcolepsy'
Status: Suspended | Type: Observational
Why Stopped: Recruitment for study has been suspended due to Covid-19.
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Ragy Tadrous, PhD Student, University of Dublin, Trinity College
Other Study IDs: Cross Sectional
Record Dates: First submitted 2020-05-12; First posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Narcolepsy; Narcolepsy 1; Narcolepsy Type 1; Narcolepsy With Cataplexy; Narcolepsy Without Cataplexy; Narcolepsy and Hypersomnia; Hypersomnolence
Keywords: Physical performance; Cardiopulmonary fitness; Muscle strength; Muscle endurance; Quality of life; Physical activity
MeSH Terms: conditions — Narcolepsy; Narcolepsy 1; Disorders of Excessive Somnolence; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Narcolepsy
  Interventions: Other: Assessment of physical performance variables

INTERVENTIONS:
Other: Assessment of physical performance variables — Other:
  Assessment of physical performance indices using the following outcome measures:
  Cardiopulmonary fitness: YMCA submaximal bike test Upper Body: ACSM press up test, Dynamometry Lower body: Wall squat test, Countermovement jump test

SUMMARY:
Narcolepsy is a sleep disorder characterised by excessive daytime sleepiness and significantly impacts quality of life. People with narcolepsy demonstrate many potential barriers to being physically active, such as sleepiness and social isolation. Very little is known about how physical performance variables may be affected and influence disease experience in people with narcolepsy. This study aims to profile the physical fitness and physical functioning variables of adults with narcolepsy and to explore the relationship between physical variables, quality of life, symptom severity and disease experience in this cohort.

DETAILED DESCRIPTION:
This study aims to profile the physical functioning variables of people with narcolepsy attending an outpatient clinic at St. James's Hospital. This will be accomplished by ascertaining the cardiopulmonary fitness, physical activity, and muscle strength and endurance of this population.

Secondary objectives of this study will be to explore the relationship between physical performance indices and sleep quality, functional ability and quality of life in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with narcolepsy type 1 or type 2 based on the International Classification of Sleep Disorders, third edition (ICSD-3) criteria for at least 6 months - diagnosis for at least 6 months will ensure that initial fluctuations due to likely starting on new drug regimen are relatively stable.
2. Eligibility screened and agreement of the participant's treating clinician in Narcolepsy out-patient clinic of St. James's Hospital that he/she can participate - to ensure that as per General Data Protection Regulation guidelines that the treating clinician eligibility screens rather than the physiotherapy study researcher.
3. Patients aged ≥18 to <65 years at the time of obtaining informed consent - as patients >18 years will not been seen in this centre, and patients >65 years may have age-related changes in cardiovascular fitness and physical activity which may be difficult to separate from those pertaining to narcolepsy diagnosis.
4. Able to understand English - as questionnaires will necessitate a sufficient level of English for completion.

Exclusion Criteria:

1. Patients with sleep disorders other than narcolepsy (e.g., moderate to severe sleep apnea syndrome, moderate to severe periodic limb movement disorder) - so results are not diluted by including conditions other than narcolepsy.
2. Any medical contraindication to exercise of moderate intensity and short duration including but not limited to cardiovascular or respiratory conditions, morbid obesity, and severe osteoarthritis of the lower extremities - as these conditions would preclude ability to conduct physical test battery.
3. Confirmed pregnancy - people with an advanced pregnancy may score differently on physical functioning/performance tests, people with a confirmed pregnancy will be excluded from study participation to limit bias.
4. Dementia or significant cognitive impairment or psychiatric illness that would preclude ability to participate in study.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The following eligibility criteria: Aged 18 to 65 years, diagnosis of type 1 or type 2 narcolepsy based on the International Classification of Sleep Disorders third edition criteria for at least six months, eligibility screened by their treating clinician, and able to understand English and follow simple instruction to enable completion of assessments. Additionally, participants will be required to provide signed and informed consent to participate in the study, and for processing of their data to be eligible for participation. Individuals with sleep disorders other than narcolepsy, contraindications to moderate-intensity exercise, confirmed pregnancy or significant psychiatric illness or cognitive impairment will be excluded from participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of oxygen uptake during cardiopulmonary exercise testing (% predicted) | 30 minutes
  The submaximal Young Men's Christian Association (YMCA) exercise test utilises the relationship between workload and heart rate to predict maximal oxygen consumption. Provides indication of cardiopulmonary fitness.
Measurement of grip strength | 15 minutes
  Objective measure of grip strength of the dominant and non-dominant hands, and will provided indication of how grip strength compares to age and gender-matched norms. Dynamometry will be used to asses muscle strength of the upper limb.
Measurement of upper limb endurance | 10 minutes
  The American College of Sports Medicine Press Up Test will be used to objectively measure muscular endurance of the upper limb. Identifies the maximum number of press ups that the participant can perform before failure.
Measurement of lower limb endurance | 10 minutes
  The wall sit test will be used to objectively measure lower limb endurance. Measures the duration a participant can maintain a wall sit until failure.
Measurement of lower limb power. | 10 minutes
  The Countermovement Jump Test will be used to objectively measure lower limb power. This test measures both jump height and peak power achieved by participants.
Measurement of physical activity | 7 days
  Actigraphy will be used to objectively measure physical activity and sedentary behaviour. Participant will be required to wear the actigraph around their waist during all waking hours except during swimming or bathing, and then send back to assessor in return-addressed envelopes.

SECONDARY OUTCOMES:
Subjective measure of Health-Related Quality of Life | 10 minutes
  Health-related quality of life will be subjectively assessed using the Short Form-36 questionnaire (Generic).
Subjective measure of Health-Related Quality of Life (sleep-disorder-specific) | 10 minutes
  Health-related quality of life will be subjectively assessed using the Functional Outcomes of Sleep Questionnaire questionnaires
Subjective measure of symptom severity | 10 minutes
  Symptom severity will be subjectively assessed through use of the Narcolepsy Severity Scale.
Subjective measure of daytime sleepiness | 5 minutes
  Daytime sleepiness will be subjectively assessed through use of the Epworth Sleepiness Scale.
Subjective measure of physical activity | 5 minutes
  Physical activity levels will be subjectively assessed through use of Physical Activity Vital Sign questionnaire.
Subjective measure of sedentary behaviour | 5 minutes
  Sedentary behaviour levels will be subjectively assessed through use of Sedentary Behaviour Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy, School of Medicine, Trinity College Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Yes
In keeping with the research policy of Trinity College Dublin, relevant and anonymised data and materials will be made available through Trinity College's Access to Research Archive (TARA) data depository.
Supporting Information: Study Protocol